CLINICAL TRIAL: NCT02106845
Title: A Phase I, Multi-center, Non-randomized, Open Label, Drug-drug-interaction Study to Determine the Effect of Multiple Doses of Regorafenib (BAY 73-4506) on the Pharmacokinetics of Probe Substrates of Transport Proteins P-gp (Digoxin; Group A) and BCRP (Rosuvastatin; Group B) in Patients With Advanced Solid Malignant Tumors
Brief Title: Effect of Regorafenib on Digoxin and Rosuvastatin in Patients With Advanced Solid Malignant Tumors.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 16674; 2013-003613-18 (EudraCT Number)
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Neoplasms
Keywords: Regorafenib; Probe substrates; Pharmacokinetics; Cancer; Safety; Advanced solid malignant tumors
MeSH Terms: conditions — Neoplasms | interventions — Digoxin; Rosuvastatin Calcium; regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- P-gp probe substrate(digoxin)+regorafenib (Experimental)
  Interventions: Drug: Digoxin; Drug: Regorafenib (Stivarga, BAY73-4506)
- Group B: BCRP probe substrate (rosuvastatin) + regorafenib (Experimental)
  Interventions: Drug: Rosuvastatin; Drug: Regorafenib (Stivarga, BAY73-4506)

INTERVENTIONS:
Drug: Digoxin — Single dose of digoxin 0.5 mg (2 tablets 0.25 mg) orally without and with regorafenib
  Arms: P-gp probe substrate(digoxin)+regorafenib
Drug: Rosuvastatin — Single dose of rosuvastatin 5mg (1 tablet 5 mg) without and with regorafenib 160 mg q.d. (4 tablets 40 mg)
  Arms: Group B: BCRP probe substrate (rosuvastatin) + regorafenib
Drug: Regorafenib (Stivarga, BAY73-4506) — Once daily orally 160 mg (4 tablets 40 mg)

SUMMARY:
Evaluate the effect of regorafenib on the pharmacokinetics of digoxin (P-gp substrate : P-glycoprotein) and rosuvastatin (BCRP substrate: Breast cancer resistant protein) by comparing their Area under time curve (AUC(0-24)) and maximum drug concentration (Cmax) on Day -7 and Cycle 1 or Cycle 2 Day 15 of regorafenib in cancer patients

ELIGIBILITY:
* Inclusion Criteria:
* The following criteria apply to ALL patients starting the study treatment:

  * Patients with histologically confirmed, locally advanced or metastatic solid tumors refractory to standard therapy or in whom regorafenib is considered a standard treatment.
  * Male or Female Caucasian patients >/= 18 years of age
  * Women of childbearing potential and men must agree to use adequate contraception before entering the program until at least 8 weeks after the last study drug administration.
  * Life expectancy of at leat 12 weeks
  * Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
  * Adequate bone marrow and liver function
  * Estimated creatinine clearance (CLcr) ≥ 30 mL/min as calculated using the Cockroft-Gault (C-G) equation.
  * Thyroid Stimulating Hormone(TSH) within normal ranges.
* The following inclusion criteria apply to Group A (digoxin + regorafenib) patients ONLY:

  * Potassium, magnesium and calcium blood levels within normal range according to the local laboratory.
* The following inclusion criteria apply to Group B (rosuvastatin + regorafenib) patients ONLY:

  * Signed genetic informed consent. Patients must be able to understand and willing to sign the written informed consent intended to screen for BCRP and OATP1B1 polymorphisms.
* Exclusion Criteria:
* For ALL patients
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days before start of study medication.
* Non-healing wound, skin ulcer, or bone fracture.
* Ongoing or active infection.
* Other anticancer treatment.
* Patients unable to swallow oral medications
* For Group A (digoxin + regorafenib):

  * Family history of sudden cardiac death.
* For Group B (rosuvastatin + regorafenib):

  * Patients with porphyria.
  * Patients with intestinal or urinary obstructions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-04-22 (Actual); Primary Completion 2015-04-27 (Actual); Study Completion 2018-06-12 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from time zero to 24 hours (AUC(0-24)) for Digoxin | On Pre-Cycle Day -7 and on Cycle 1 Day15 or Cycle 2 Day 15
Maximum drug concentration (Cmax) in plasma for Digoxin | On Pre-Cycle Day -7 and on Cycle 1 Day15 or Cycle 2 Day 15
Area under the plasma concentration-time curve from time zero to 24 hours (AUC(0-24)) for rosuvastatin | On Pre-Cycle Day -7 and on Cycle 1 Day15 or Cycle 2 Day 15
Maximum drug concentration (Cmax) in plasma for rosuvastatin | On Pre-Cycle Day -7 and on Cycle 1 Day15 or Cycle 2 Day 15

SECONDARY OUTCOMES:
Tumor Response following RECIST criteria | From first dose up to 3 months after end of treatment
Number of participants with adverse events as a measure of safety and tolerability | Up to 30 days after last dose
Number of participants with drug related adverse events as a measure of safety and tolerability | Up to 30 days after last dose

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (4):
- Germany (3):
  - Freiburg im Breisgau, Baden-Wurttemberg
  - Frankfurt am Main, Hesse
  - Herne, North Rhine-Westphalia
- Budapest, Hungary